CLINICAL TRIAL: NCT01693952
Title: Sepsis in Neutropenic Patients: Autologous Stem Cell Transplantation as Model: a Transcriptomic Approach.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00322-41; 2012-08 (Other: AP HM)
Record Dates: First submitted 2012-05-21; First posted 2012-09-26 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Sepsis in Neutropenic Patients
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- blood samples (Experimental)
  Interventions: Biological: blood draw

INTERVENTIONS:
Biological: blood draw

SUMMARY:
Treatment of cancer, and more particularly of haematological malignancies, partly relies on chemotherapy. Most therapeutic regimens display various toxicities, one of the most common being haematological toxicity, affecting the three lineages. While anaemia and thrombopenia can be overcome by haematological growth factors and transfusion, one of the most severe life-threatening toxicity is sepsis that develops during neutropenia. Neutropenia, despite the use of granulocyte colony-stimulating factors (G-CSF) and antibiotics, is still a major limitation in chemotherapy which is responsible for the majority of treatment-related morbidity and mortality and for prolonged hospitalisation.

In neutropenic patients, sepsis is more frequent and more severe than in non-neutropenic patients. While the occurence of neutropenia and sepsis is often unpredictable and thus difficult to study in a prospective way, stem cell transplantation represents a quite convenient model to study such a question. Autologous stem cell transplantation indications in haematology are mainly multiple myeloma and relapsed lymphoma or Hodgkin disease. Briefly, after a mobilization procedure, a graft of patient's hematopoietic stem cells is collected by cytapheresis and frozen. When the patient has reached complete remission by conventional chemotherapy, he benefits from a very high dose myeloablative chemotherapy (called "conditioning regimen"). The "conditioning regimen" targeted to have high antitumoral activity leads to a "cytokine storm" resulting in a "programmed inflammation". 36 hours after the lasting of the conditioning regimen, the CD34+ cells are thawed and infused to the patient. Thus neutropenia usually begins at D4 post transplantation and lasts for 10 days, until graft becomes "functional". Thus, the timing and duration of neutropenia are very homogeneous. During neutropenia, fever and sepsis are very frequent (>80% patients), thus, most patient will be informative regarding sepsis, and there is an easy possibility of biological sampling before" programmed inflammation" (due to conditioning regimen), after inflammation before sepsis, then during and after the sepsis. Since the patient is hospitalized, the kinetic monitoring is quite easy

ELIGIBILITY:
Inclusion Criteria:

* the criteria required to be candidate in an ASCH in our service(department) (age 18 - 66 years, myélome in 1 ° in reply partial line or lymphoma or complete answer after one 2 ° line, absence of preliminary visceral failure).

Informed, willing patients and having given their agreement in writing.

Exclusion Criteria:

* Refusal of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
blood samples | 3 YEARS
  transcriptomic profile identification

SECONDARY OUTCOMES:
blood samples | 3 YEARS
  the observed profile in patients developing fever and sepsis in comparison with patients not developing such complications
blood samples | 3 YEARS
  the prediction, for each patient, a transcriptomic signature linked to a higher risk developing a sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France